CLINICAL TRIAL: NCT06867432
Title: Efficacy and Safety of Yttrium-90 Microspheres Selective Internal Radiotherapy Combined with Immune Checkpoint Inhibitors and Anti-angiogenesis Drugs Sequential Hepatic Arterial Infusion Chemotherapy (HAIC) for Hepatocellular Carcinoma
Brief Title: Efficacy and Safety of Yttrium-90 Microspheres Selective Internal Radiotherapy Combined with Immune Checkpoint Inhibitors and Anti-angiogenesis Drugs Sequential HAIC for Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, HuiKai Li, Chief Physician, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC-2025-0003
Record Dates: First submitted 2025-02-24; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SIRT-Y90+HAIC+PD-1 or PD-L1 inhibitors +targeted therapy (Experimental): Yttrium (90Y) -SIRT treatment: SIRT enables resin-based yttrium (90Y) microspheres. The radioactivity of yttrium (90Y) and the therapeutic dose were calculated by the body surface product method. The designated dose of yttrium (90Y) microsphere injection was infused after hepatic arterial catheterization, tumor donor artery. The treatment sessions targeted the liver lobe with a larger tumor volume.
  Patients were monitored for 2 days after treatment. In cases of local tumor progression and contraindications, SIRT may be repeated. Hepatic arterial infusion chemotherapy: specific drug dose, drug method according to current guidelines and drug marketing instructions. Every 3 weeks starting after 3 weeks of yttrium (90Y) -SIRT. PD-L1/PD-1 inhibitors and targeted therapy as specified in the guidelines are allowed to be administered during each treatment
  Interventions: Drug: Combination Product：t: SIRT-Y90 +HAIC+Atezolizumab + Bevacizumab

INTERVENTIONS:
Drug: Combination Product：t: SIRT-Y90 +HAIC+Atezolizumab + Bevacizumab — Single or two-staged delivery of SIRT-Y90 (4 to 6 weeks), followed by 1200mg atezolizumab + 15mg/kg bevacizumab administered by IV at every 3 weeks for 18 months.
  HAIC：administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks.

SUMMARY:
To observe and evaluate the efficacy and safety of selective internal radiotherapy (SIRT) based on transarterial radioembolization with yttrium (90Y) microspheres combined with immune checkpoint inhibitors and anti-angiogenic-drug sequential hepatic arterial infusion chemotherapy (HAIC) for the treatment of initially unresectable hepatocellular carcinoma with transformation potential.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 and ≤75 years of age, regardless of gender;
* Hepatocellular carcinoma (HCC) diagnosed clinically or pathologically with the following characteristics and assessed by the investigator to be initially not amenable to surgical resection but with the potential for surgical resection after conversion therapy;
* The tumour is confined to a unilateral hepatic lobe, with no extrahepatic metastases and no clinical evidence of high pressure on the imperial vein;
* CNLC stage Ib-IIIa;
* ECOG PS score: 0-1;
* At least one measurable lesion according to mRECIST criteria;
* Child-Pugh A;
* For patients with active hepatitis B virus (HBV): HBV-DNA must be <2,000 IU/mL and must have received at least 14 days of anti-HBV treatment (based on current guidelines, e.g., entecavir) prior to the start of study treatment and be willing to receive antiviral treatment for the full duration of the study; HCV-RNA-positive patients must receive antiviral treatment according to guidelines; and HCV-RNA-positive patients must receive antiviral treatment according to guidelines. HCV-RNA-positive patients must be receiving antiviral therapy according to guidelines and have liver function within CTCAE class 1 ascending;
* No severe fluid, renal, or coagulation dysfunction:

  1. Gynecological examination (excluding the use of any gynecological fluid component and cell growth within 14 days) 1) Neutrophil count (NE) >1.5 x 109/L; 2) Glucose count (NE) >1.5 x 109/L; 3) Glucose count (NE) >1.5 x 109/L; 2) Hemoglobin count (HGB) >90 g/L; 3) Platelet count (PLT) >75×109/L;
  2. Liver and kidney function:

  <!-- -->

  1. Serum creatinine ≤2.0×ULN;
  2. Total bilirubin (TBIL) ≤ 2.0 × ULN;
  3. Aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 × ULN;
* Completion of 99mTc-MAA and SPECT/CT to meet the treatment requirements for 90Y-SIRT, including but not limited to: (1) pulmonary shunt fraction <20%; (2) single pulmonary absorbed dose <25Gy or cumulative pulmonary absorbed dose <30Gy (Twice Y90 Treatment interval 4-6 weeks);
* An expected life expectancy of ≥3 months;
* No previous treatment with transhepatic arterial embolisation (TAE, cTACE or D-TACE), targeted therapy, immunotherapy, radiotherapy or pellet implantation, or SIRT;
* Women of childbearing potential must have a negative pregnancy test (serum) or urine HCG test within 7 days prior to enrolment and be willing to use appropriate contraception during the trial and for 8 weeks after the last dose of the test drug; for men, they should be surgically sterilised or agree to use appropriate contraception during the trial and for 8 weeks after the last dose of the test drug;
* The patients were willing to enter the study and signed an informed consent form.

Exclusion Criteria:

* Known fibroplaque HCC, hydatidiform HCC, or mixed hepatocellular carcinoma;
* Refractory ascites (despite optimal diuretic therapy) or any other clinical signs of liver failure;
* Untreated or incompletely treated hydronephrosis and/or fundal varices or those at high risk of bleeding as assessed by the investigator, or a history of bleeding due to hydronephrosis or fundal varices within 1 month prior to entry;
* Major surgical treatment or chemotherapy, radiotherapy or other systemic treatment of the lesion within 1 month prior to entry;
* Previous allogeneic nickel-hydride cell or solid organ transplantation;
* Active autoimmune disease requiring systemic therapy (use of palliative medications, steroids, or immunosuppressants); or Thymosin-α1, etc.) within 30 days of the study.
* Have received a live attenuated vaccine within 4 weeks prior to the study, or expect to receive such a vaccine during treatment or within 5 months of the last dose.
* Uncontrolled medical conditions including, but not limited to, persistent infections (other than viral hepatitis), symptomatic cardiac failure, unstable heartburn, colic, cardiac arrest, and heartburn.Uncontrolled medical conditions include, but are not limited to, persistent infections (except viral hepatitis), symptomatic cardiac failure, unstable cardiac colic, irregular heartbeat or severe mental illness;
* Uncontrolled high blood pressure (systolic > 150 mmHg and/or diastolic > 100 mmHg). 10. other active malignant tumours;
* Other active malignancies (completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder cancer).Other active malignancies (except completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, and superficial bladder carcinoma, and any other cancer that has not recurred for at least 5 years);
* A history of allergy to therapeutic agents and compounds of similar composition;
* Contraindications to study drug or SIRT therapy, or to angiography as assessed by the Investigator;
* Pregnant or lactating women and those planning to conceive;
* Have participated in other research studies in the last 3 months;
* Inability to understand or unwillingness to sign a written informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR mRESIST | Prior to surgery
  from the date of enrollment to death from any cause.

SECONDARY OUTCOMES:
Transformation success rate | Up to approximately 48 months
  Defined as having at the same time: 1) R0 resection can be achieved and sufficient residual liver volume (FLR) can be preserved; 2) Child-Pugh A or B; 3) ECOG PS score 0 - 1;(4) There is no tumour thrombosis in the main internal secretion vein or inferior vena cava. (5)No tumour thrombus in the main and inferior vena cava; 5) No contraindication to hepatectomy;
R0 Resection Rate | Up to approximately 48 months
  R0 resection rate (proportion of resected participants obtaining an R0 resection). R0 resection is defined as a microscopically margin-negative resection, in which no tumor (gross or microscopic) remains in the primary tumor bed.
Progression-free survival (PFS) | Up to approximately 48 months
  The time from randomization to the date of tumor progression at any site in the body or death from any cause, whichever is earlier. For those who remain alive and have not progressed, PFS will be censored on the date of the last evaluable tumor assessment on or before the time of analysis or the end of study treatment, whichever is earlier.
Overall survival (OS) | Randomization to death from any cause (up to approximately 3 years)
  OS is defined as the time from randomization to death from any cause.
Pathologic Complete Response (pCR) Rate | Up to approximately 48 months
  pCR rate is defined as the proportion of participants with an absence of residual tumor at the time of surgery, as assessed by central pathological review.

IPD SHARING:
Plan to Share IPD: No